CLINICAL TRIAL: NCT06439732
Title: Impact of Using an Hemodynamic Monitoring System on Anesthetic Consumption During Abdominal Surgery
Acronym: HERMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, RUSSO ANDREA, principal investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6704
Record Dates: First submitted 2024-05-22; First posted 2024-06-03 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Hypotension During Surgery
Keywords: Anestethic comsumption; hemodynamic monitoring

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): In this group we will use a continuous non-invasive hemodynamic monitoring system (Acumen IQ cuff)
  Interventions: Device: Acumen IQ cuff
- Control (No Intervention): In this group we will use the oscillometric non-invasive blood pressure monitoring system

INTERVENTIONS:
Device: Acumen IQ cuff — Use of Acumen IQ cuff for haemodynamic monitoring
  Arms: Intervention

SUMMARY:
In this study investigators will study the association between the use of an hemodynamic monitoring system and the anesthetic consumption in patients following major abdominal surgery. Investigators will randomise patients for a control group and an intervention group. Patients belonging to intervention group will be monitored with a non-invasively continue system (Acumen IQ cuff sensor), while the control group will be monitored with a non-invasive intermittent pressure system. The total amount of mL of Sevoflurane will be registered in both groups and the difference will be considered as the aim of our study

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* signature of informed medical consent

Exclusion Criteria:

* BMI> 30
* eGFR<30
* NYHA III-IV
* severe cardiac valvular diseases
* absence of informed medical consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Reduction in Anesthetic consumption | During surgery

SECONDARY OUTCOMES:
number hypotensive episodes | during surgery
duration hypotensive episodes | during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Russo, MD, Principal Investigator — Fondazione Policlinico universitario Agostino Gemelli
Locations (1):
- Fondazione Policlinico Universitario "A. Gemelli" IRCCS, Roma, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided